CLINICAL TRIAL: NCT02059915
Title: An Open-Label, Randomized, 2-Cohort, Single-Dose, Crossover Study Of 40 Mg Doses Of Pf-00345439 To Evaluate The Bioequivalence Of Modified Formulation K Vs. Original Formulation X Under Intermediate-Fat Fed Conditions And To Estimate Relative Bioavailability Under Fasting Conditions In Healthy Volunteers
Brief Title: Single-Dose, Crossover Study To Compare Bioavailability Of Two Formulations Under Fed And Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501015
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: pharmacokinetics; bioequivalence; bioavailability; oxycodone
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment B (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment C (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment D (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation X, single dose, under fed conditions
  Arms: Treatment A
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, under fed conditions
  Arms: Treatment B
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation X, single dose, under fasting conditions
  Arms: Treatment C
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, under fasting conditions
  Arms: Treatment D

SUMMARY:
To Compare The Bioavailability Of 40 Mg Doses Of Pf-00345439 Modified Formulation K Vs. Original Formulation X Under Fed And Fasting Conditions In Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 18 and 55 years of age

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Positive urine drug test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Concentration at time 24 hours (C24) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Plasma Decay Half-Life (t1/2) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Saint Paul, Minnesota, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501015&StudyName=Single-Dose%2C%20Crossover%20Study%20To%20Compare%20Bioavailability%20Of%20Two%20Formulations%20Under%20Fed%20And%20Fasted%20Conditions